CLINICAL TRIAL: NCT02418949
Title: Altering Activation Patterns in the Distal Upper Extremity After Stroke
Brief Title: Altering Activation Patterns Post-stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Elliot Roth, Medical Director, Patient Recovery Unit, Attending Physician, RIC Professor & Chairman, PM&R, Northwestern Feinberg School of Medicine, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00078099; 1R01HD075813-01A1 (NIH)
Record Dates: First submitted 2015-02-05; First posted 2015-04-17 (Estimated); Results first posted 2021-07-13 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Stroke; Muscle Spasticity; Hemiparesis
Keywords: hand; rehabilitation; active movement training; passive cyclical stretching
MeSH Terms: conditions — Stroke; Muscle Spasticity; Paresis | interventions — Cyproheptadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cyproheptadine + AMP (Experimental): Cyproheptadine will be titrated up to the chronic dose prior to involvement in hand therapy.
  Week 1 dose: 4mg taken twice daily (orally) Week 2 dose: 8mg taken twice daily (orally) Week 3 dose: (chronic dose): 8 mg taken three times daily (orally). Chronic dose will be maintained throughout the 6 weeks of Active movement practice (AMP) treatment (1 hour sessions 3x/week). Dose will be titrated down to zero in the 2 weeks following treatment.
  Interventions: Drug: Cyproheptadine; Other: Active Movement Practice (AMP)
- Placebo for Cyproheptadine + Stretching (Placebo Comparator): Placebo for Cyproheptadine will be titrated up to the chronic dose prior to involvement in hand therapy.
  Week 1 dose: 4mg taken twice daily (orally) Week 2 dose: 8mg taken twice daily (orally) Week 3 dose: (chronic dose): 8 mg taken three times daily (orally). Chronic dose will be maintained throughout the 6 weeks of passive cyclical stretching treatment (1 hour sessions 3x/week). Each session will involve 20 min of stretching followed by 10 minutes of rest.
  Dose will be titrated down to zero in the 2 weeks following treatment.
  Interventions: Drug: Placebo for Cyproheptadine; Other: Passive Cyclical Stretching
- Cyproheptadine + Stretching (Active Comparator): Cyproheptadine will be titrated up to the chronic dose prior to involvement in hand therapy.
  Week 1 dose: 4mg taken twice daily (orally) Week 2 dose: 8mg taken twice daily (orally) Week 3 dose: (chronic dose): 8 mg taken three times daily (orally). Chronic dose will be maintained throughout the 6 weeks of passive cyclical stretching treatment (1 hour sessions 3x/week). Each session will involve 20 min of stretching followed by 10 minutes of rest.
  Dose will be titrated down to zero in the 2 weeks following treatment.
  Interventions: Drug: Cyproheptadine; Other: Passive Cyclical Stretching
- Placebo for Cyproheptadine + AMP (Active Comparator): Placebo for Cyproheptadine will be titrated up to the chronic dose prior to involvement in hand therapy.
  Week 1 dose: 4mg taken twice daily (orally) Week 2 dose: 8mg taken twice daily (orally) Week 3 dose: (chronic dose): 8 mg taken three times daily (orally). Chronic dose will be maintained throughout the 6 weeks of Active movement practice (AMP) treatment (1 hour sessions 3x/week). Dose will be titrated down to zero in the 2 weeks following treatment.
  Interventions: Drug: Placebo for Cyproheptadine; Other: Active Movement Practice (AMP)

INTERVENTIONS:
Drug: Cyproheptadine — Cyproheptadine will be titrated up to the chronic dose prior to involvement in hand therapy as well as gradually down to zero in the two weeks following treatment.
  Week 1 dose: 4mg taken twice daily (orally) Week 2 dose: 8mg taken twice daily (orally) Week 3 dose: (chronic dose): 8 mg taken three times daily (orally). Week 4-9: (chronic dose): 8 mg taken three times daily (orally). Week 10: 8 mg taken twice daily (orally). Week 11: 4 mg taken twice daily (orally). Week 12: no drug
  Other Names: cyproheptadine hydrochloride USP; cyproheptadine HCl; Periactin
  Arms: Cyproheptadine + AMP; Cyproheptadine + Stretching
Drug: Placebo for Cyproheptadine — Cyproheptadine will be titrated up to the chronic dose prior to involvement in hand therapy as well as gradually down to zero in the two weeks following treatment.
  Week 1 dose: 4mg taken twice daily (orally) Week 2 dose: 8mg taken twice daily (orally) Week 3 dose: (chronic dose): 8 mg taken three times daily (orally). Week 4-9: (chronic dose): 8 mg taken three times daily (orally). Week 10: 8 mg taken twice daily (orally). Week 11: 4 mg taken twice daily (orally). Week 12: no drug
  Other Names: placebo
  Arms: Placebo for Cyproheptadine + AMP; Placebo for Cyproheptadine + Stretching
Other: Active Movement Practice (AMP) — Participants will alternate between active training with a custom video game and a robot active-assistive Voice and EMG-Driven Actuated (VAEDA) glove during active training occupational therapy.
  Arms: Cyproheptadine + AMP; Placebo for Cyproheptadine + AMP
Other: Passive Cyclical Stretching — Participants will wear the actuated device/glove for the duration of the training sessions (2 20-min stints followed by 10 min of rest) during which time the actuated glove will cyclically stretch the joints of the digits in the hand between flexion and extension while remaining passive/relaxed.
  Arms: Cyproheptadine + Stretching; Placebo for Cyproheptadine + Stretching

SUMMARY:
This study evaluates a new rehabilitation approach for stroke survivors in the chronic phase of recovery in which the combination of drug therapy (cyproheptadine) and active movement practice (AMP) is used to encourage increased voluntary muscle control and strength.

DETAILED DESCRIPTION:
In this four arm parallel design you will be randomly assigned to one of 4 groups:

Group 1) cyproheptadine and active movement therapy, Group 2) placebo and active movement therapy, Group 3) cyproheptadine and passive stretching, or Group 4) placebo and passive stretching.

The groups will be blinded so neither you nor the research staff (or even the study doctor) will know which drug (Cyproheptadine or placebo) you receive. Only the RIC pharmacist will have access to this information until all participants complete the entire study. Although you and the research staff administering the training sessions will know if you have been assigned to the active movement practice (AMP) or passive cyclical stretching group, it is important not to discuss this information with the rater (evaluator) or the study doctor.

Cyproheptadine is an anti-serotonergic and anti spastic agent. It is expected to reduce the unwanted muscle hyper excitability (one measure of spasticity) common after stroke.

During the course of the treatment you will be required to make several visits per week to RIC to either be evaluated or participate in the treatment sessions. Evaluations last approximately 2 hours and will be performed at the beginning of weeks 1, 2, 3 and 4, during the middle of treatment (beginning of week 7), at the end of training (beginning of week 10) as well as a final follow-up visit one month after the end of treatment (beginning of week 14). The training sessions will occur from weeks 4 through week 9 and will involve 1.5-hr. sessions (1 hr training plus setup time) 3 times per week.

The investigators hypothesize that the group receiving the combined cyproheptadine and active movement therapy will have better outcomes than the groups receiving cyproheptadine or active movement therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Chronic, severe hand hemiparesis resulting from a single stroke (Chedoke- McMaster Stroke Assessment: Stage of Hand 2 or 3)
* Single stroke occurring at least 6 months prior to enrollment
* Spasticity
* Capacity to provide informed consent

Exclusion Criteria:

* Excessive pain in paretic upper limb
* Hemispatial neglect (as assessed by the Behavioral Inattention Test)
* Apraxia (as assessed by the FABERS battery)
* Botulinum toxin injection in the upper extremity within the past 6 months
* Introduction of new anti-spasticity medication within the past 6 months
* Orthopaedic impairments
* History of seizure disorder
* Other major health impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-11; Primary Completion 2019-08 (Actual); Study Completion 2023-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Derek G Kamper, PhD, Study Director — North Carolina State University; Elliot Roth, MD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ochoa JM, Listenberger M, Kamper DG, Lee SW. Use of an electromyographically driven hand orthosis for training after stroke. IEEE Int Conf Rehabil Robot. 2011;2011:5975382. doi: 10.1109/ICORR.2011.5975382. PMID 22275586
- [Background] Ochoa J, Dev Narasimhan YJ, Kamper DG. Development of a portable actuated orthotic glove to facilitate gross extension of the digits for therapeutic training after stroke. Annu Int Conf IEEE Eng Med Biol Soc. 2009;2009:6918-21. doi: 10.1109/IEMBS.2009.5333630. PMID 19964456
- [Background] Thielbar KO, Triandafilou KM, Fischer HC, O'Toole JM, Corrigan ML, Ochoa JM, Stoykov ME, Kamper DG. Benefits of Using a Voice and EMG-Driven Actuated Glove to Support Occupational Therapy for Stroke Survivors. IEEE Trans Neural Syst Rehabil Eng. 2017 Mar;25(3):297-305. doi: 10.1109/TNSRE.2016.2569070. Epub 2016 May 17. PMID 27214905
- [Derived] Kamper D, Barry A, Bansal N, Stoykov ME, Triandafilou K, Vidakovic L, Seo N, Roth E. Use of cyproheptadine hydrochloride (HCl) to reduce neuromuscular hypertonicity in stroke survivors: A Randomized Trial: Reducing Hypertonicity in Stroke. J Stroke Cerebrovasc Dis. 2022 Oct;31(10):106724. doi: 10.1016/j.jstrokecerebrovasdis.2022.106724. Epub 2022 Aug 30. PMID 36054974
- [Derived] Barry AJ, Triandafilou KM, Stoykov ME, Bansal N, Roth EJ, Kamper DG. Survivors of Chronic Stroke Experience Continued Impairment of Dexterity But Not Strength in the Nonparetic Upper Limb. Arch Phys Med Rehabil. 2020 Jul;101(7):1170-1175. doi: 10.1016/j.apmr.2020.01.018. Epub 2020 Feb 28. PMID 32113974

RESULTS

PARTICIPANT FLOW:
Groups:
- Cyproheptadine + AMP: Cyproheptadine will be titrated up to the chronic dose prior to involvement in hand therapy.
  Week 1 dose: 4mg taken twice daily (orally) Week 2 dose: 8mg taken twice daily (orally) Week 3 dose: (chronic dose): 8 mg taken three times daily (orally). Chronic dose will be maintained throughout the 6 weeks of Active movement practice (AMP) treatment (1 hour sessions 3x/week). Dose will be titrated down to zero in the 2 weeks following treatment.
  Cyproheptadine: Cyproheptadine will be titrated up to the chronic dose prior to involvement in hand therapy as well as gradually down to zero in the two weeks following treatment.
  Week 1 dose: 4mg taken twice daily (orally) Week 2 dose: 8mg taken twice daily (orally) Week 3 dose: (chronic dose): 8 mg taken three times daily (orally). Week 4-9: (chronic dose): 8 mg taken three times daily (orally). Week 10: 8 mg taken twice daily (orally). Week 11: 4 mg taken twice daily (orally). Week 12: no drug
  Active Movement Practice (AMP): Participants will alternate between active training with a custom video game and a robot active-assistive Voice and EMG-Driven Actuated (VAEDA) glove during active training occupational therapy.
- Placebo for Cyproheptadine + Stretching: Placebo for Cyproheptadine will be titrated up to the chronic dose prior to involvement in hand therapy.
  Week 1 dose: 4mg taken twice daily (orally) Week 2 dose: 8mg taken twice daily (orally) Week 3 dose: (chronic dose): 8 mg taken three times daily (orally). Chronic dose will be maintained throughout the 6 weeks of passive cyclical stretching treatment (1 hour sessions 3x/week). Each session will involve 20 min of stretching followed by 10 minutes of rest.
  Dose will be titrated down to zero in the 2 weeks following treatment.
  Placebo for Cyproheptadine: Cyproheptadine will be titrated up to the chronic dose prior to involvement in hand therapy as well as gradually down to zero in the two weeks following treatment.
  Week 1 dose: 4mg taken twice daily (orally) Week 2 dose: 8mg taken twice daily (orally) Week 3 dose: (chronic dose): 8 mg taken three times daily (orally). Week 4-9: (chronic dose): 8 mg taken three times daily (orally). Week 10: 8 mg taken twice daily (orally). Week 11: 4 mg taken twice daily (orally). Week 12: no drug
  Passive Cyclical Stretching: Participants will wear the actuated device/glove for the duration of the training sessions (2 20-min stints followed by 10 min of rest) during which time the actuated glove will cyclically stretch the joints of the digits in the hand between flexion and extension while remaining passive/relaxed.
- Cyproheptadine + Stretching: Cyproheptadine will be titrated up to the chronic dose prior to involvement in hand therapy.
  Week 1 dose: 4mg taken twice daily (orally) Week 2 dose: 8mg taken twice daily (orally) Week 3 dose: (chronic dose): 8 mg taken three times daily (orally). Chronic dose will be maintained throughout the 6 weeks of passive cyclical stretching treatment (1 hour sessions 3x/week). Each session will involve 20 min of stretching followed by 10 minutes of rest.
  Dose will be titrated down to zero in the 2 weeks following treatment.
  Cyproheptadine: Cyproheptadine will be titrated up to the chronic dose prior to involvement in hand therapy as well as gradually down to zero in the two weeks following treatment.
  Week 1 dose: 4mg taken twice daily (orally) Week 2 dose: 8mg taken twice daily (orally) Week 3 dose: (chronic dose): 8 mg taken three times daily (orally). Week 4-9: (chronic dose): 8 mg taken three times daily (orally). Week 10: 8 mg taken twice daily (orally). Week 11: 4 mg taken twice daily (orally). Week 12: no drug
  Passive Cyclical Stretching: Participants will wear the actuated device/glove for the duration of the training sessions (2 20-min stints followed by 10 min of rest) during which time the actuated glove will cyclically stretch the joints of the digits in the hand between flexion and extension while remaining passive/relaxed.
- Placebo for Cyproheptadine + AMP: Placebo for Cyproheptadine will be titrated up to the chronic dose prior to involvement in hand therapy.
  Week 1 dose: 4mg taken twice daily (orally) Week 2 dose: 8mg taken twice daily (orally) Week 3 dose: (chronic dose): 8 mg taken three times daily (orally). Chronic dose will be maintained throughout the 6 weeks of Active movement practice (AMP) treatment (1 hour sessions 3x/week). Dose will be titrated down to zero in the 2 weeks following treatment.
  Placebo for Cyproheptadine: Cyproheptadine will be titrated up to the chronic dose prior to involvement in hand therapy as well as gradually down to zero in the two weeks following treatment.
  Week 1 dose: 4mg taken twice daily (orally) Week 2 dose: 8mg taken twice daily (orally) Week 3 dose: (chronic dose): 8 mg taken three times daily (orally). Week 4-9: (chronic dose): 8 mg taken three times daily (orally). Week 10: 8 mg taken twice daily (orally). Week 11: 4 mg taken twice daily (orally). Week 12: no drug
  Active Movement Practice (AMP): Participants will alternate between active training with a custom video game and a robot active-assistive Voice and EMG-Driven Actuated (VAEDA) glove during active training occupational therapy.
Period: Overall Study
Arm/Group | Cyproheptadine + AMP | Placebo for Cyproheptadine + Stretching | Cyproheptadine + Stretching | Placebo for Cyproheptadine + AMP
Started | 23 | 22 | 26 | 25
Completed | 20 | 21 | 23 | 24
Not Completed | 3 | 1 | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: 1 Participant in "Cyproheptadine + AMP" & 1 Participant in "Cyproheptadine + Stretching" did not continue past enrollment to baseline assessment
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyproheptadine + AMP | Placebo for Cyproheptadine + Stretching | Cyproheptadine + Stretching | Placebo for Cyproheptadine + AMP | Total
Number analyzed (Participants) | 22 | 22 | 25 | 25 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (8.1) | 57.1 (11.2) | 58.9 (13.1) | 57.3 (9.5) | 58.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 10 | 8 | 35
  Male | 14 | 13 | 15 | 17 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 21 | 23 | 23 | 68
  Not Hispanic or Latino | 21 | 1 | 2 | 2 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 2 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 11 | 9 | 12 | 13 | 45
  White | 8 | 13 | 11 | 11 | 43
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Chedoke McMaster Scale of Hand [Count of Participants; unit: Participants] — The Chedoke McMaster Stroke Assessment is comprised of 6 impairment inventories, which can be administered individually. Hand Impairment is scored on a 7-point scale with each point corresponding to seven stages of motor recovery. Higher scores indicate better motor recovery post-stroke. Stage 2 is indicated as spasticity presented as resistance to passive movement. Stage 3 shows marked spasticity but with voluntary movement of the fingers.
  Participants
    Equal or less than 2 | 6 | 11 | 6 | 8 | 31
    Equal or Greater than 3 | 16 | 11 | 19 | 17 | 63
Fugl-Meyer Upper Extremity Assessment [Mean (Standard Deviation); unit: Score] — The Fugl-Meyer (FM) Assessment of Motor Recovery evaluates and measures recovery in post-stroke hemiplegic patients. The FM uses a 3-point ordinal scale from 0 (cannot perform) to 2 (performs fully). The FM has 5 domains with a maximum score of 226 points. Subscales can be administered with out using the full FM. The Upper Extremity component consists of 33 items with a score range of 0-66. A higher score indicates better performance.
  Score | 15 (8.1) | 12.9 (5.5) | 16.1 (7.1) | 15.6 (5.6) | 15 (6.6)
Lesion Side [Count of Participants; unit: Participants]
  Left | 10 | 7 | 11 | 12 | 40
  Right | 12 | 15 | 14 | 13 | 54
Time Since Stroke onset (Years) [Mean (Standard Deviation); unit: years] | 5.9 (4.3) | 5.4 (5.3) | 5.6 (4.7) | 8.5 (8.6) | 6.4 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Completion Time for Graded Wolf Motor Function Test (GWMFT)
Description: GWMFT is a clinical outcome measure comprised of 15 timed tasks focusing on upper extremity function. Maximum allowable time per task is 120 seconds.
Time Frame: baseline and 9 weeks (immediately post intervention)
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Cyproheptadine + AMP | Placebo for Cyproheptadine + Stretching | Cyproheptadine + Stretching | Placebo for Cyproheptadine + AMP
Number analyzed (Participants) | 20 | 21 | 23 | 24
Seconds | -3.66 [-7.95 to 0.63] | -0.51 [-3.62 to 2.60] | -4.00 [-7.72 to -0.28] | -3.89 [-8.65 to 0.88]

2. Secondary Outcome: Change in Grip Relaxation Time (Following a Maximum Voluntary Contraction (MVC)
Description: Following a maximum voluntary contraction (MVC) -- Time (s) required for muscle electromyographic (EMG) signals to reduce to within 3 SD of pre-MVC EMG activity.
Time Frame: baseline and 9 weeks (immediately post intervention)
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Cyproheptadine + AMP | Placebo for Cyproheptadine + Stretching | Cyproheptadine + Stretching | Placebo for Cyproheptadine + AMP
Number analyzed (Participants) | 20 | 21 | 23 | 24
Seconds | -1.66 [-2.79 to 0.54] | -0.96 [-3.20 to 1.28] | -1.06 [-3.19 to 1.07] | -2.65 [-4.70 to -0.59]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during study enrollment, from screening to the final follow up appointment (13 total weeks after initial screening)
Arm/Group | Cyproheptadine + AMP | Placebo for Cyproheptadine + Stretching | Cyproheptadine + Stretching | Placebo for Cyproheptadine + AMP
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22 | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/23 | 2/22 | 1/26 | 0/25
Other Adverse Events (participants affected / at risk) | 19/23 | 15/22 | 18/26 | 21/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyproheptadine + AMP (N=23) | Placebo for Cyproheptadine + Stretching (N=22) | Cyproheptadine + Stretching (N=26) | Placebo for Cyproheptadine + AMP (N=25)
Convulsions (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHF Exacerbation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary Blockage (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot Wound (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyproheptadine + AMP (N=23) | Placebo for Cyproheptadine + Stretching (N=22) | Cyproheptadine + Stretching (N=26) | Placebo for Cyproheptadine + AMP (N=25)
Dry Mouth (General disorders) | 9 (9) | 9 (9) | 11 (11) | 9 (9)
Low Energy (General disorders) | 10 (10) | 7 (7) | 12 (12) | 4 (4)
Weight Gain (Metabolism and nutrition disorders) | 7 (7) | 6 (6) | 9 (9) | 5 (5)
Low Motivation (Psychiatric disorders) | 1 (1) | 5 (5) | 9 (9) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (6) | 5 (5) | 6 (6) | 6 (6)
Restless/Jittery (General disorders) | 4 (4) | 3 (3) | 4 (4) | 3 (3)
Slowness/Trouble getting moving (General disorders) | 3 (3) | 6 (6) | 7 (7) | 5 (5)
Frequent Urination (Renal and urinary disorders) | 7 (7) | 6 (6) | 7 (7) | 4 (4)
Sleep Problems (General disorders) | 3 (3) | 4 (4) | 5 (5) | 5 (5)
Difficulty Urinating (Renal and urinary disorders) | 4 (4) | 2 (2) | 2 (2) | 2 (2)
Memory Problems (General disorders) | 2 (2) | 8 (8) | 9 (9) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT02418949/Prot_000.pdf
  • Statistical Analysis Plan (2014-06-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT02418949/SAP_001.pdf
  • Informed Consent Form (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT02418949/ICF_002.pdf